CLINICAL TRIAL: NCT07012460
Title: Pulsed Field Ablation for Cavotricuspid Isthmus Dependent Atrial Flutter Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Prof, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pulse CTI study
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Cavotricuspid Isthmus Dependent Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTI ablation (Other): CTI ablation will be performed with PFA. Coronary angiogram will be performed at baseline in LAO 45 degree before and after each set of ablations. The CTI block will be rechecked with 3D mapping system and multipolar catheter. If there is persistent CTI conduction, ablation will be repeated until CTI block is achieved. If CTI block cannot be achieved with repeated PFA ablation, ablation with radiofrequency will be allowed to achieve block. Patient will come back for follow up at 3 months for a remapping procedure. During the remapping procedure, a RCA coronary angiogram will be performed to exclude late coronary damage.
  Interventions: Device: CTI ablation

INTERVENTIONS:
Device: CTI ablation — CTI ablation will be performed with PFA. Before ablation, The RA geometry will be created with a multipolar catheter. Coronary angiogram will be performed at baseline in LAO 45 degree before and after each set of ablations. After ablation, a 15-minute waiting period will be mandated. The CTI block will be rechecked with 3D mapping system and multipolar catheter. If there is persistent CTI conduction, ablation will be repeated until CTI block is achieved. This will be followed by another 15 minutes of waiting period before rechecking the block across CTI, and so on. TNG will be prepared. It will be given via intracoronary route in 100-200mcg bolus if severe spasm is observed. If CTI block cannot be achieved with repeated PFA ablation, ablation with radiofrequency will be allowed to achieve block. Patient will come back for follow up at 3 months for a remapping procedure. During the remapping procedure, a RCA coronary angiogram will be performed to exclude late coronary damage.

SUMMARY:
Pulsed field ablation (PFA) has been demonstrated to be safe and effective in achieving pulmonary vein isolation in patients with atrial fibrillation (AF). Coexisting atrial flutter is common in patients with AF. It is therefore appealing to treat the atrial futters with PFA. The use of PFA for extra-pulmonary ablation, such as linear ablation at the mitral or cavo-tricuspid isthmus (CTI) has been investigated. When PFA is applied near a coronary vessel, acute coronary spasm is a common observation, which has been reported to be reversible and largely mitigated by pre-emptive intravenous or intracoronary nitroglycerine (TNG) injection. A recent clinical study based on qualitative coronary angiogram reported no apparent coronary stenosis 6 months after PFA. However, quantitative measurements were not provided. While acute conduction block is easy to create with pulsed field ablation catheters, the long-term lesion durability is unknown. The circular array pulsed field ablation catheter was shown to be safe and effective in achieving pulmonary vein isolation. This study aims to evaluate the safety and efficacy of pulsed-field ablation for CTI flutters.

This study will be a multicenter prospective cohort study involving 30 patients undergoing ablation for atrial fibrillation and CTI flutter. The decision for ablation will be a clinical decision based on existing class I and II guideline recommendations.

The atrial fibrillation ablation procedure will be performed as per routine clinical practice. Procedure will be performed with a 3-D electro-anatomical system guidance. Pulmonary vein isolation (PVI) will be performed with pulsed field ablation with a circular array catheter (Pulse Select system, Medtronic). After confirming PVI, extrapulmonary ablation will be performed per clinically need. CTI ablation will be performed with PFA as planned.

Patient will be managed by usual clinical care after ablation. They will come back for follow up at 3 months for a remapping procedure. During the remapping procedure, a RCA coronary angiogram will be performed to exclude late coronary damage. A multipolar catheter will be inserted via right femoral vein to check for conduction block across CTI. If there is ongoing conduction, a repeat ablation will be performed with radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrial fibrillation who are clinically planned to undergo AF ablation and atrial flutter ablation per guideline recommendations

Exclusion Criteria:

1. >80 years old or <18 years old
2. Known severe coronary artery disease
3. Prior history of atrial flutter or atrial fibrillation ablation
4. Refusal for remapping or coronary angiogram
5. Contraindication for coronary angiogram
6. Pregnancy
7. Expected life expectancy <1 year
8. Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of residual conduction | In 3 months follow up
  Evaluate rate of residual conduction across CTI in 3-month remapping
Rate of coronary artery damage | In 3 months follow up
  Evaluate rate of coronary artery damage in 3-month repeat coronary angiogram
Rate of acute severe coronary spasm | In 3 months follow up
  Evaluate rate of acute severe coronary spasm induced by PFA (>70% diameter reduction or ST change)

SECONDARY OUTCOMES:
Rate of clinical recurrence of atrial arrhythmia | In 3 months follow up
  Evaluate rate of clinical recurrence of atrial arrhythmia at 3 months
Number of PFA applications | In ablation procedure
  Evaluate number of PFA applications required to achieve CTI block
Rate of successful acute conduction block by PFA alone | In ablation procedure
  Evaluate rate of successful acute conduction block by PFA alone
Rate of successful acute conduction block in all patients (with PFA or PFA + RFA) | In ablation procedure
  Evaluate rate of successful acute conduction block in all patients (with PFA or PFA + RFA)
Number of mapping points in right atrium in electroanatomic system | In mapping procedure
  Evaluate number of mapping points in right atrium in electroanatomic system

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong